CLINICAL TRIAL: NCT03021954
Title: The Role of Platelet Rich Plasma in Supporting the Recovery of Post-partum Levator Ani Muscle Trauma
Brief Title: Platelet Rich Plasma in Levator Ani Muscle Trauma
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Dr Cipto Mangunkusumo General Hospital (Other)
Collaborators: Indonesia University (Other)
Responsible Party: Principal Investigator, Fernandi Moegni, M.D., Obstetric and gynaecologist, Urogynaecologist, Dr Cipto Mangunkusumo General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: DCiptoMGHFMoegni
Record Dates: First submitted 2017-01-11; First posted 2017-01-16 (Estimated); Results first posted 2024-01-29 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2023-07

CONDITIONS: Pelvic Floor Disorders
Keywords: platelet rich plasma; levator ani muscle; post-partum trauma; ballooning trauma; levator ani muscle strength
MeSH Terms: conditions — Pelvic Floor Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention Group (Experimental): Platelet rich plasma injected intramuscularly in pelvic floor muscle immediately following labor and before perineoraphy, simultaneously with the injection of local anesthesia
  Interventions: Biological: Platelet Rich Plasma
- Control Group (No Intervention): No intervention given, patient will only get local anesthesia injection before perineoraphy

INTERVENTIONS:
Biological: Platelet Rich Plasma — Platelet rich plasma is an autologous blood with high amount of platelet. It produced by obtaining patient's whole blood and processed by centrifugation and activation by CaCl2.
  Other Names: PRP
  Arms: Intervention Group

SUMMARY:
Levator trauma (ballooning) often occurs after vaginal delivery. Platelet rich plasma injection after delivery showed reduced hiatal area and maintain levator muscle strength.

DETAILED DESCRIPTION:
This study aims to see if PRP has a beneficial effect on the repair of pelvic floor muscle damage in primipara. Therefore, this single-blinded randomized clinical trial compares the pelvic floor muscle repair in primipara following labor between the interventional group who received intramuscular PRP injection in levator ani muscle and the control group, as assessed by ultrasonography, perineometry. The ultrasonography outcome measures include lower hiatal area during Valsalva. The assessments are performed at multiple time points, which are before labor, 24-48 hours post-labor, 40 days post-labor, and 3 months post-labor.

ELIGIBILITY:
Inclusion Criteria:

* primigravida, in third trimester pregnancy
* plan to do vaginal birth
* have a clear address and telephone number that can be contacted
* consent to participate in this study

Exclusion Criteria:

* history of pelvic floor disorder before pregnancy
* history of pelvic surgery
* avulsion of levator ani muscle (seen in USG)
* unstable hemodynamic
* trombocytopenia (< 150,000)
* anemia (Hb< 10)
* sepsis
* infection on perineum
* corticosteroid intake within last 2 weeks
* smoking
* hematopoetic or bone cancer
* delivery by c-section
* no perineoraphy after birth

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 116 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2019-01 (Actual); Study Completion 2020-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fernandi Moegni, MD,OBGYN(C), Principal Investigator — FKUI/RSCM
Locations (1):
- Primary Care Centre, Jakarta Pusat, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study started in November 2016 until July 2019. We included all women who had a vaginal delivery in public health center (Puskesmas), and several referral hospitals. Minimal sampel size calculated for this study was 23 subjects each group, with 20 % additional for anticipating loss to follow up subjects. Therefore, minimal sample size was 29 each group.
Pre-assignment Details: We obtained 116 primigravid women. Fifty-three subjects were drop-out failed to finish the study. Five subjects were excluded from the study cause were detected having avulsion (macro trauma) injury at 40 days post-partum evaluation that was considered as severe degree of trauma and would made bias to the healing process. Finally, there were 58 subjects who successfully followed the examination until the end of the study.
Groups:
- Platelet Rich Plasma: as many as 29 subjects were included in the intervention group. All of the subjects underwent PRP injection at levator ani muscle directly after vaginal delivery. Afterward, all of the subjects returned to control at 40 days post-partum for pelvic ultrasound examination assessing levator hiatal area and perineometry examination for assessing levator ani muscle strength. Then, the subject was asked to return at 3 months post-partum to perform a similar examination.
- Lidocaine (Placebo): as many as 29 subjects were included in the control group. All of the subjects underwent lidocaine 1% (placebo) injection at levator ani muscle directly after vaginal delivery. Afterward, all of the subjects returned to control at 40 days post-partum for pelvic ultrasound examination assessing levator hiatal area and perineometry examination for assessing levator ani muscle strength. Then, the subject was asked to return at 3 months post-partum to perform a similar examination.
Period: Overall Study
Arm/Group | Platelet Rich Plasma | Lidocaine (Placebo)
Started | 43 | 73 (We excluded 43 subjects due to lost to follow-up, one subject had levator ani muscle avulsion. Therefore only 29 subjects in the control group finished all the examinations in this study.)
Completed | 29 | 29
Not Completed | 14 | 44
Not completed — Lost to Follow-up | 10 | 43
Not completed — Subjects had avulsion trauma | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Intervention: The intervention group receive a single dose of PRP that was produced from their own blood. We injected the PRP in the levator ani muscle when we did the perineorrhaphy procedure.
  A baseline measurement was taken at the third trimester of pregnancy (when they come to do antenatal control). Then, we do a follow-up assessment at 40 weeks and three months post-partum.
- Control: The control group only receive lidocaine (placebo) when we did the perineorrhaphy procedure.
  A baseline measurement was taken at the third trimester of pregnancy (when they come to do antenatal control). Then, we do a follow-up assessment at 40 weeks and three months post-partum.
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 29 | 29 | 58
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 30.5 [24.5 to 36.5] | 25 [20 to 30] | 28.5 [22 to 34.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 29 | 58
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 29 | 29 | 58
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Levator Hiatal Area at Valsalva [Median (Inter-Quartile Range); unit: cm2] | 20.64 [12.9 to 28.38] | 20.35 [14.78 to 25.94] | 20.37 [13.5 to 27.24]
Levator ani muscle strength [Mean (Standard Deviation); unit: cmH2O] | 37.45 (13.89) | 41.45 (18.05) | 39.39 (16.09)
Baby birth weight [Median (Inter-Quartile Range); unit: gram] | 3042 [2606 to 3478] | 3100 [2640 to 3560] | 3100 [2639 to 3561]

OUTCOME MEASURES:

1. Primary Outcome: Changes of Levator Hiatal Area During Valsava
Description: Changes in lower hiatal area during valsalva in various measurements (compared to baseline value), measured using translabial 3D ultrasound. With the translabial technique at an angle of 70 degrees or more, the entire levator hiatus and surrounding muscles (pubococcygeus and puborectalis) can be visualized. It is hoped that ultrasound is more reproducible because axial measurements are easier with minimal dimensional images, at rest, valsalva, or contraction.
Time Frame: Baseline (third trimester), 40 days post-partum, 3 months post-partum
Measure: Median (Inter-Quartile Range); unit: Cm2
Groups:
- Intervention: All intervention subjects underwent pelvic ultrasound examination for assessing levator hiatal area during valsalva at antenatal visit (baseline), 40 days post-partum, 3 months post-partum
- Control: All control subjects underwent pelvic ultrasound examination for assessing levator hiatal area during valsalva at antenatal visit, 40 days post-partum, 3 months post-partum
Arm/Group | Intervention | Control
Number analyzed (Participants) | 29 | 29
Cm2
  Pre-intervention | 20.64 [12.9 to 28.38] | 20.35 [14.78 to 25.92]
  40 days post-partum | 22.35 [18.4 to 26.3] | 21.41 [15.14 to 27.68]
  3 months post-partum | 17.57 [11.92 to 23.22] | 18.54 [9.56 to 27.5]
Statistical Analysis 1: Comparison: Intervention vs Control; The null hypothesis is in the intervention group, we expect a decrease in the area of the levator hiatus at 40 days and 3 months post-partum. Power 90 % confidence interval β = 0.10, α = 0.05; Test type: Superiority; p = 0.086, Wilcoxon (Mann-Whitney)

2. Primary Outcome: Changes in Pelvic Floor Muscle Contraction
Description: Changes in pelvic floor muscle contraction in various measurements (compared to baseline), measured using perineometer
Time Frame: Baseline (third trimester), 40 days post partum, and 3 months post partum
Measure: Mean (Standard Deviation); unit: CmH2O
Groups:
- Intervention: All intervention subjects underwent levator ani muscle strength examination using perineometer at antenatal / third trimester, at 40 days post-partum, at 3 months post-partum
- Control: All control subjects underwent levator ani muscle strength examination using perineometer at antenatal / third trimester, at 40 days post-partum, at 3 months post-partum
Arm/Group | Intervention | Control
Number analyzed (Participants) | 29 | 29
CmH2O
  Pre-Intervention | 37.45 (13.89) | 41.45 (18.05)
  40 days post-partum | 28.94 (16.49) | 28.79 (15.86)
  3 months post-partum | 35.84 (18.81) | 30.88 (18.33)
Statistical Analysis 1: Comparison: Intervention vs Control; The null hypothesis is platelet rich plasma can maintain or increase levator ani muscle contractions post-partum; Test type: Equivalence; p = 0.29, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: 3 months
Description: The intervention procedure in this study is platelet rich plasma injection at levator ani muscle during the during perineorraphy after childbirth which is a normal procedure of labor. Treatment was carried out according to the post-partum care protocol, so incidence of infection can be avoided.
Groups:
- Intervention: We collect adverse events by asking the subject and physical examination (especially site of injection)
- Control: No different collection method with the intervention group
Arm/Group | Intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/29
Other Adverse Events (participants affected / at risk) | 0/29 | 0/29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2018-01-15): https://cdn.clinicaltrials.gov/large-docs/54/NCT03021954/Prot_000.pdf
  • Statistical Analysis Plan (2018-01-15): https://cdn.clinicaltrials.gov/large-docs/54/NCT03021954/SAP_001.pdf
  • Informed Consent Form (2018-01-15): https://cdn.clinicaltrials.gov/large-docs/54/NCT03021954/ICF_002.pdf